CLINICAL TRIAL: NCT04840537
Title: Comparison of Two Diagnostic Strategies in Indeterminate Biliary Stenosis: Exploration by Retrograde Cholangioscopy From the Outset or After Failure of Conventional Techniques
Brief Title: Cholangioscopy or Conventional Techniques for Indeterminate Biliary Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frederic PRAT, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Frederic PRAT, MD, PhD, Principal Investagator, Medical Doctor, Hôpital Cochin
Organization: Hôpital Cochin (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SFED 131
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Malignant Biliary Stenosis
Keywords: biliary stenosis; cholangioscopy; cholangiocarcinoma; ERCP
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cytological brushing followed by cholangioscopy in case of failure (Active Comparator)
  Interventions: Procedure: endoscopic retrograde cholangiopancreatography with cholangioscopy in the first procedure of ERCP
- cholangioscopy from the start (Experimental)
  Interventions: Procedure: endoscopic retrograde cholangiopancreatography with cholangioscopy in the first procedure of ERCP

INTERVENTIONS:
Procedure: endoscopic retrograde cholangiopancreatography with cholangioscopy in the first procedure of ERCP — endoscopic retrograde cholangiopancreatography with cholangioscopy in the first procedure for exploration of an indeterminate biliary stenosis and biliary drainage

SUMMARY:
Biliary stenosis not associated with a mass is difficult to diagnose with certainty. The diagnosis is usually based on a first-line cytological study of biliary brushing, which allows a diagnosis in 30 to 50% of cases. In the event of negativity, it is then possible to perform a cholangioscopy in a second step, which allows better sensitivity by performing biopsies. Performing cholangioscopy from the start could potentially save time and avoid disturbances associated with intermediate biliary stenting.

The main objective is to compare two strategies for exploring indeterminate biliary stenosis (1st vs. 2nd line retrograde cholangioscopy) in terms of diagnostic performance. The secondary objectives are to compare the same two strategies in terms of effectiveness, side effects and cost-effectiveness.

The primary outcome measure is the diagnostic yield (performance) of the initial investigation of indeterminate biliary stenosis: cytological brushing followed by cholangioscopy in case of failure (control group) or cholangioscopy from the start (study group).

ELIGIBILITY:
Inclusion Criteria:

* Presence of intra- or extrahepatic biliary stenosis, involving the main bile ducts: common hepatic duct, right and left hepatic ducts
* Presence of clinical jaundice and / or biological cholestasis (GGT> 3N)
* Absence of visible mass near the biliary stenosis after initial morphological assessment by abdominal CT scan, MRI with biliary sequences.
* Endoscopic ultrasound performed and not having allowed the acquisition of material of diagnostic interest by guided puncture of the lesion.
* No history of ERCP in the 6 months preceding inclusion and no biliary prosthesis (plastic or metal) in place at the time of inclusion
* Collegial validation of the need for a formal diagnosis of indeterminate biliary stenosis in order to guide therapeutic management
* Patients aged 18 to 85
* Patient who gave his consent to participate in the study
* No contraindication to anesthesia (ASA 1, 2,3)
* Patient affiliated to a social security scheme (beneficiary or beneficiary)
* Absence of pregnancy and current contraception in women of childbearing age

Exclusion Criteria:

* Presence of a manifest tissue mass in relation to the biliary stenosis on CT and / or MRI imaging.
* Very strong presumption of the etiological diagnosis of biliary stenosis given the history (history, background): i.e. liver surgery, cholecystectomy, autoimmunity
* History of ERCP and / or percutaneous biliary drainage in the 6 months preceding inclusion
* Presence of a plastic or metal biliary prosthesis in place at the time of inclusion
* History of cephalic duodeno-pancreatectomy or hepatico-jejunal anastomosis
* Non-passable stenosis of the main bile duct
* Severe coagulopathy, thrombocytopenia <75,000 G / L, treatment with clopidogrel cannot be interrupted even temporarily
* Anesthetic contraindication (ASA 4)
* Inability to obtain informed consent
* person deprived of liberty

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-12-26 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2022-12-26 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield (performance) of the initial investigation of indeterminate biliary stenosis: cytological brushing followed by cholangioscopy in case of failure (control group) or cholangioscopy from the start (study group). | 48 months
  Diagnostic performance is expressed primarily by sensitivity for the diagnosis of malignancy.

SECONDARY OUTCOMES:
Specific rate of diagnosis with cholangioscopy by spyglass used in 1st or 2nd intention | 48 months
Rate of adverse events related to diagnostic procedures in each of the 2 groups | 48 months
Comparison of the costs of the 2 diagnostic strategies | 48 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Beaujon, Clichy, France

IPD SHARING:
Plan to Share IPD: No